CLINICAL TRIAL: NCT01646112
Title: Living in Lynch Syndrome Limbo: Exploring the Meaning of Uncertain Genetic Test Results
Brief Title: Uncertain Genetic Test Results for Lynch Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912126; 12-HG-N126
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-02-05

CONDITIONS: HNPCC
Keywords: Uncertainty; HNPCC; Lynch Syndrome; Genetic Tests
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

* Individuals have varying tolerances for receiving ambiguous information. However, not much is known about how ambiguous genetic testing information is received. Also, not much is known about how at-risk individuals internalize and process these results. More information is needed about how this information affects a person s life.
* Lynch Syndrome is a genetic condition that carries a high risk of colon cancer and other cancers. Individuals at risk for Lynch Syndrome can have genetic testing for it. The test may confirm a diagnosis and determine actions that can be taken. Results from genetic testing can also affect the perspectives of relatives who might also be affected. However, genetic testing can also produce variants of unknown significance (VUS). VUS are data that may not provide enough information to make decisions. Researchers want to study people who have received a VUS result for genetic testing for Lynch Syndrome.

Objectives:

- To learn more about the impact and experience of receiving a VUS for Lynch Syndrome genetic testing.

Eligibility:

- Individuals at least 18 years of age who have recently had a VUS result on a genetic test for Lynch Syndrome.

Design:

* Participants will be asked to answer demographic questions. They will also have a 45- to 60-minute phone interview.
* During the phone interview, participants will be asked a series of questions about their diagnosis. They will be asked about how they received the result and how they felt right after receiving it. They will also discuss who they have spoken to about the result.

DETAILED DESCRIPTION:
In the field of cancer genetics, clinicians and patients have encountered challenges related to the significance of unclassified genetic variants (UV) or variants of unknown significance (VUS). As the field of medical genetics moves toward whole genome sequencing (WGS), these challenges will inevitably become more frequent. VUS represent ambiguous and uncertain data, for which pathogenicity has not been demonstrated or excluded in published literature, mutation databases or on the basis of other clinical findings. Such variants present a clinical interpretation challenge and also evoke new counseling dilemmas for the understanding and psychosocial impact of uncertain genetic test results. This exploratory study aims to seek insight into the psychological impact of receiving a VUS through semi-structured interviews with 30 to 40 individuals who have received a VUS test result for one of the Lynch Syndrome/Hereditary Nonpolyposis Colorectal Cancer (HNPCC) mismatch repair genes. The interviews will focus on the experience of receiving this result and any cognitive, affective or behavioral effects related to the uncertainty of the result. Interviews will be transcribed and subjected to thematic analysis to identify themes running through the interviews. Understanding the impact of receiving a VUS may identify areas for future intervention studies to minimize negative effects of these events. Additionally, these data may contribute to the formulation of guidelines surrounding the consent for and disclosure of VUS s for other diseases and ultimately for WGS.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Individuals who have received a VUS for Lynch Syndrome must be over 18, have telephone access and speak English. Individuals will be excluded if they ve received their results less than 3 months earlier or more than 6 years ago.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04-25; Study Completion 2016-02-05

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Antoniou A, Pharoah PD, Narod S, Risch HA, Eyfjord JE, Hopper JL, Loman N, Olsson H, Johannsson O, Borg A, Pasini B, Radice P, Manoukian S, Eccles DM, Tang N, Olah E, Anton-Culver H, Warner E, Lubinski J, Gronwald J, Gorski B, Tulinius H, Thorlacius S, Eerola H, Nevanlinna H, Syrjakoski K, Kallioniemi OP, Thompson D, Evans C, Peto J, Lalloo F, Evans DG, Easton DF. Average risks of breast and ovarian cancer associated with BRCA1 or BRCA2 mutations detected in case Series unselected for family history: a combined analysis of 22 studies. Am J Hum Genet. 2003 May;72(5):1117-30. doi: 10.1086/375033. Epub 2003 Apr 3. PMID 12677558
- [Background] Kresse A, Jacobowitz DM, Skofitsch G. Distribution of calcitonin gene-related peptide in the central nervous system of the rat by immunocytochemistry and in situ hybridization histochemistry. Ann N Y Acad Sci. 1992 Jun 30;657:455-7. doi: 10.1111/j.1749-6632.1992.tb22798.x. No abstract available. PMID 1637098
- [Background] Boks DE, Trujillo AP, Voogd AC, Morreau H, Kenter GG, Vasen HF. Survival analysis of endometrial carcinoma associated with hereditary nonpolyposis colorectal cancer. Int J Cancer. 2002 Nov 10;102(2):198-200. doi: 10.1002/ijc.10667. PMID 12385019